CLINICAL TRIAL: NCT06367842
Title: Contribution of Systematic Pathological Examination of Orthopaedic Specimens to the Early Diagnosis of Tranthyretin Amyloid Heart Disease
Brief Title: Orthopaedic Specimen Pathology and Early Diagnosis of ATTR Cardiopathy (ATTR-ORTHO)
Acronym: ATTR-ORTHO
Status: Recruiting | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: MED-02-2023
Record Dates: First submitted 2024-03-06; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: ATTR Amyloidosis; Cardiopathy; Carpal Tunnel Syndrome; Lumbar Spine Stenosis; Hip Prosthesis; Knee Prosthesis
Keywords: ATTR amyloidosis; cardiac amyloidosis; orthopaedic surgery
MeSH Terms: conditions — Heart Diseases; Carpal Tunnel Syndrome; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the frequency of ATTR amyloid, cardiac involvement and associated features, in 150 patients aged 50 or more years, and operated for an idiopathic carpal tunnel syndrome, lumbar spine stenosis or total hip or knee arthroplasty for primary osteoarthritis. The main questions to be answered are:

1. What is the frequency of ATTR deposits in samples retrieved during surgery?
2. What is the frequency of cardiac involvement in ATTR positive patients?
3. What are the preoperative predictors of ATTR deposits? Participants will

   * have operative samples stained by Congo red in search of amyloid, which will be typed by immunochemistry in positive samples,
   * undergo a multimodal imaging search for cardiac involvement, if ATTR is identified,
   * undergo a preoperative complete clinical examination, including collection of medical history, ECG, biochemical tests, and imaging (ultrasound scans of rotator cuff and hip capsule in all participating patients, of the carpal tunnel in patients operated at this site, and MRI + standing profile radiography of the lumbar spine, in patients operated for lumbar stenosis)
   * ATTR positive patients will be proposed to be followed-up by a reference center, with the aim of an early diagnosis of cardiac involvement, allowing efficient mamagement.

Researchers will assess the frequency of ATTR deposits at each operated site, the frequency or ATTR cardiopathy in ATTR + patients, and will compare demographic, clinical, biochemical, and imaging features in patients with and without ATTR deposits, to guide the indications of pathological examination during these frequent orthopedic surgeries

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 50 or over
2. having signed an informed consent form
3. undergoing surgery for

   1. idiopathic carpal tunnel syndrome
   2. or lumbar spinal canal stenosis
   3. or prosthetic replacement of a hip or knee for primary osteoarthritis

Exclusion Criteria:

1. secondary carpal tunnel syndrome (inflammatory rheumatism, diabetes, hypothyroidism, etc.)
2. Indication of prosthesis for a condition other than primary osteoarthritis.
3. Known amyloidosis
4. Refusal of consent
5. Inability to understand the study
6. Age < 50 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the inclusion criteria in a single orthopaedic surgery center located in Paris, France
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
frequency of ATTR amyloidosis | 18 months
  presence of ATTR amyloidosis in surgical samples by immunohistochemistry performed when samples countain amyloi by Congo red.ATTR will be semiquantitalively assessed using a published scale.

SECONDARY OUTCOMES:
presence of ATTR cardiopathy | 20 months
  Diagnosis by multimodal imaging(bone scintigraphy, cardiac US scan, MRI)
proportion of wild type and hereditary ATTR | 20 months
  hereditary: patients exibit a mutation of the TTR gene, wild type: no mutation. TTR genotyping will determine if the gene is muted (hereditary ATTR) or not (wild type).
Description of preoperative predictors of ATTR | 18 months
  features more frequent in patients diagnosed with ATTR versus not:
  - demographic and clinical characteristics,
  will be collected before surgery and compared in ATTR positive and ATTR negative patients.
Description of preoperative predictors of ATTR | 18 months
  features more frequent in patients diagnosed with ATTR versus not:
  - imaging characteristics (USscans of rotator cuff, hip capsula and carpal tunel)
  will be collected before surgery and compared in ATTR positive and ATTR negative patients.
preoperative predictors of ATTR | 18 months
  biochemical features more frequent in patients diagnosed with ATTR versus not:
  * troponine (g/L)
  * BNP (ng/L)
  * proteuniria (ng/L) will be collected before surgery and compared in ATTR positive and ATTR negative patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Mutualist Montsouris Institute, Paris, France